CLINICAL TRIAL: NCT06312202
Title: Fatal and Non-fatal Drowning Incidents in Danish Harbours: a Nationwide Registry-based Study Using the Danish Prehospital Drowning Data From 2016-2023
Brief Title: Drowning Incidents in Danish Harbours
Acronym: DROWN_HARBOR
Status: Not yet recruiting | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Principal Investigator, Prehospital Center, Region Zealand
Other Study IDs: DROWN_HARBOUR
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Drowning; Drown; Drowning; Anoxia; Drowning, Near; Drowning; Asphyxia; Drowning and Nonfatal Submersion; Drowning or Immersion of Unknown Intent; Drowning and Submersion, Undetermined Intent; Drowning and Submersion While in Natural Water; Drowning and Submersion Due to Sailboat Sinking; Drowning and Submersion Due to Fall Off Ship
Keywords: Danish Drowning Formula; Danish Prehospital Drowning Data; Denmark; Registry; Database; Cohort; Drowning; Harbour; Emergency Medical Service; Submersion
MeSH Terms: conditions — Drowning; Hypoxia; Near Drowning; Asphyxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fatal drowning: This group of patients experienced a drowning incident defined as the process of experiencing respiratory impairment from submersion or immersion in liquid and died within 30 days after the incident as a consequence of the submersion injury.
  Interventions: Other: Drowning
- Non-fatal drowning: This group of patients experienced a drowning incident defined as the process of experiencing respiratory impairment from submersion or immersion in liquid and survived until 30 days after the incident.
  Interventions: Other: Drowning

INTERVENTIONS:
Other: Drowning — Drowning is defined as the process of experiencing respiratory impairment from submersion or immersion in liquid.

SUMMARY:
A recent study reported significantly increased mortality from drowning-related out-of-hospital cardiac arrest in Danish harbours compared to other public places (e.g., public pools, coastlines, and lakes). Accurate and reliable data are necessary before establishing specific educational, preventative, rescue, or treatment strategies to reduce the number of drowning incidents in Danish harbours and improve survival. Therefore, it is essential to characterise drowning incidents in Danish harbours and analyse risk factors associated with fatal drowning.

DETAILED DESCRIPTION:
Based on the GPS coordinates and advanced text-searching, it is possible to identify drowning incidents in Danish harbours and extract data from the Danish Prehospital Drowning Data.

This study is a nationwide registry-based study with data from the Danish Prehospital Drowning Data from 2016 to 2023. In this study, we will use 30-day mortality to differentiate between fatal and non-fatal drowning.

The primary objective is to estimate the yearly incidence of fatal and non-fatal drowning incidents in Danish harbours treated by the EMS from 2016 to 2023 and calculate the fatal to non-fatal ratio. The secondary objective is to assess risk factors associated with 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* All the patients registered in the Danish Prehospital Drowning Data from 2016-2023 will be assessed for inclusion AND
* Incidents registered at GPS coordinates corresponding to a Danish harbour OR
* Incidents identified using advanced text-search algorithm searching for "harbour"-related words

Exclusion Criteria:

* Patients without a 30-day follow-up (e.g., due to missing or invalid civil registration numbers) and patients with a valid DNAR code will be excluded from the mortality analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target condition in this study is drowning, irrespective of follow-up at 30 days (fatal or non-fatal). We used the WHO definition of drowning supported by the clarification statement for non-fatal drowning as the case definition to identify drowning (target condition) during the manual validation.
  The study unit is the individual drowning patient. The target population are all fatal and non-fatal drowning patients in Danish harbours treated by the EMS in Denmark since 2016. Due to the comprehensive search criteria in the Danish Drowning Formula, it is reasonable to believe that the target population is identical to the study population.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Yearly incidence of drowning incidents | 30 days after the drowning incident
  Yearly incidence of fatal and non-fatal drowning incidents in Danish harbours treated by the EMS from 2016-2023
Fatal to non-fatal drowning ratio | 30 days after the drowning incident
  Cumulated counts of fatal to non-fatal drowning incidents from 2016-2023

SECONDARY OUTCOMES:
Assess risk factors associated with 30-day mortality | 30 days after the drowning incident
  Hypothesis-driven assessment of risk factors associated with drowning-related 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Helle Collatz Christensen, MD, PhD, Study Director — pre
Locations (1):
- Prehospital Center, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
The datasets used and analysed during the current study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Breindahl N, Wolthers SA, Jensen TW, Holgersen MG, Blomberg SNF, Steinmetz J, Christensen HC; Danish Cardiac Arrest Group. Danish Drowning Formula for identification of out-of-hospital cardiac arrest from drowning. Am J Emerg Med. 2023 Nov;73:55-62. doi: 10.1016/j.ajem.2023.08.024. Epub 2023 Aug 15. PMID 37619443